CLINICAL TRIAL: NCT04747886
Title: Supplementing Evidence-based Commercial Weight Management Program With Inhibitory Control Training: a Pilot Study
Brief Title: Inhibitory Control Adult Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Sarah Salvy, Professor, Department of Medicine, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001164
Record Dates: First submitted 2021-01-25; First posted 2021-02-10 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WW Only (Active Comparator): Participants will receive 3-month access to the WW digital program.
  Interventions: Behavioral: WW Only
- WW + PolyRules! (Experimental): Participants will receive 3-month access to the WW digital program and the PolyRules! app.
  Interventions: Behavioral: WW + PolyRules!

INTERVENTIONS:
Behavioral: WW Only — WW is a structured behavioral weight management program that focuses on diet, physical activity and mindset skills. The dietary approach is based on creating an energy deficit diet to produce weight loss while also being attentive to the quality of the calories. Specifically, the WW program assigns SmartPoints values to foods based on calories, sugar, saturated fat and protein. In addition, particular foods are assigned a points value of zero (0) to encourage a healthier eating pattern (e.g. fruits, vegetables, non-fat yogurt, fish).
  Arms: WW Only
Behavioral: WW + PolyRules! — In addition to WW, participants will be asked to engage in daily cognitive training using the PolyRules! app for three months. They will be instructed to start with 20-min of daily cognitive training and to progressively increase their training time to 30-min.
  Arms: WW + PolyRules!

SUMMARY:
The purpose of this pilot study is to explore the benefits of supplementing the WW (formerly Weight Watchers) online program with a cognitive training game (PolyRules!) among adults with overweight or obesity.

DETAILED DESCRIPTION:
This two-arm pilot study will be used to estimate the effect size in weight loss of supplementing the WW (formerly Weight Watchers) online program with gamified inhibitory control training (PolyRules!) among adults with overweight or obesity. Participants ages 18 and older (n=30) will be randomly assigned to one of two study arms: (1) WW (formerly Weight Watchers) only or (2) WW + Gamified inhibitory control training (PolyRules!). All participants will complete demographic, medical history questionnaires and cognitive assessment battery at baseline/enrollment and after completing the 3-month intervention protocol. All interactions with PolyRules! and WW will be passively recorded to monitor the frequency of interaction with WW and PolyRules!.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Read, write and speak English with acceptable visual acuity
* BMI between 25-40 kg/m^2

Exclusion Criteria:

* Currently enrolled in weight loss interventions or undergoing bariatric surgery
* Pregnant women
* Individuals with severe cognitive delays or visual/hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah-Jeanne Salvy, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Pacific Design Center, West Hollywood, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WW Only | WW + PolyRules!
Started | 14 | 20
Completed | 13 | 16
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 4

BASELINE CHARACTERISTICS:
Population: WW Only included 13 participants who contributed baseline data. WW + PolyRules! included 17 participants who contributed baseline data, one participant in this group withdrew after providing baseline data but before completing the intervention and providing post-intervention data for a final analytic sample of 29.
Groups:
- Total: Total of all reporting groups
Arm/Group | WW Only | WW + PolyRules! | Total
Number analyzed (Participants) | 13 | 17 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (10.0) | 51.9 (13.4) | 49.5 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 16 | 26
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 9 | 14 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 17 | 30
BMI [Mean (Standard Deviation); unit: kg/m^2] | 35.1 (6.6) | 35.3 (6.3) | 35.2 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: BMI at Three Months
Description: BMI will be calculated by aggregating participants' self-reported height in meters and weight in kilograms at baseline and at 3 months. Throughout the study, participants will be asked to self-report their weight through the WW (formerly Weight Watchers) online app. This data will be used to calculate change in BMI.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | WW Only | WW + PolyRules!
Number analyzed (Participants) | 13 | 16
kg/m^2 | 34.53 (6.5) | 34.43 (6.2)

2. Other Pre Specified Outcome: Change in Visuo-spatial Working Memory Based on Performance on the Corsi Task.
Description: Change in visuo-spatial working memory will be assessed by participant's performance on the Corsi tasks. Performance will be measured by assessing the number of correct sequences, such that a larger number of correct sequences is a more favorable outcomes.
Time Frame: Baseline, 3 months
Reporting Status: Not Posted, anticipated posting 2025-01

3. Other Pre Specified Outcome: Change in Performance on the Letter-number Task.
Description: Change in working memory will also be assessed using participant's performance on the letter-number task. Performance will be measured by looking at error rates, such that higher error rates are worse outcomes.
Time Frame: Baseline, 3 months
Reporting Status: Not Posted, anticipated posting 2025-01

4. Other Pre Specified Outcome: Change in Performance on the N-back Task.
Description: Change in working memory will be assessed using participant's performance on the N-back task. Performance will be measured by looking at the number of errors such that more errors is a worse outcome.
Time Frame: Baseline, 3 months
Reporting Status: Not Posted, anticipated posting 2025-01

5. Other Pre Specified Outcome: Change in Performance on the Cancellation Task.
Description: Attention and inhibitory control will be assessed using participant's change in performance on the cancellation task. Performance will be measured by summing up the total number of errors committed within a specific time frame, such that lower scores are more favorable.
Time Frame: Baseline, 3 months
Reporting Status: Not Posted, anticipated posting 2025-01

6. Other Pre Specified Outcome: To Explore Whether Inhibitory Control Training Confers Any Increases in Self-reported Physical Activity.
Description: Physical activity will be assessed using participant's self-reported physical activity levels through the WW (formerly Weight Watchers) online app. This data will be leveraged to assess changes in engagement in energy balance behaviors by capturing information on the type, duration and intensity of activity.
Time Frame: Baseline, 3 months
Reporting Status: Not Posted, anticipated posting 2025-01

7. Other Pre Specified Outcome: Change in Performance on the Countermanding Task.
Description: Attention and inhibitory control will also be assessed using participant's change in performance on the countermanding task. Performance will be measured by summing the number of accurate responses within a 15 second timeframe, such that higher scores are more favorable.
Time Frame: Baseline, 3 months
Reporting Status: Not Posted, anticipated posting 2025-01

8. Other Pre Specified Outcome: To Explore Whether Inhibitory Control Training Confers Any Benefits in Self-reported Diet
Description: Diet quality will be assessed using participant's self-reported food intake through the WW (formerly Weight Watchers) online app. This data will be leveraged to assess changes in adherence to dietary guidelines for fruits and vegetables, servings of whole grains, red/processed meats, alcoholic beverages and food/beverages with added sugars.
Time Frame: Baseline, 3 months
Reporting Status: Not Posted, anticipated posting 2025-01

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of each participant's consent until the active intervention (12 weeks) and end of study procedures were completed, totaling 14-16 weeks.
Description: N=34 enrolled, and n=3 withdrew prior to baseline. Participants are monitored for adverse events until they withdrew, were lost to follow up, or completed the study. WW Arm: n=13 monitored until end of study completion. WW + Poly! Arm: n=18 enrolled, and n=2 dropped out before study completion.
Arm/Group | WW Only | WW + PolyRules!
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/18
Other Adverse Events (participants affected / at risk) | 0/13 | 0/18

LIMITATIONS AND CAVEATS:
1. Small and homogeneous sample of participants. Individuals who took part in the study were highly educated, affluent and 86.7% were women.
2. Short intervention duration compared to other weight management trials.
3. Reliance on self-report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT04747886/Prot_SAP_ICF_000.pdf